CLINICAL TRIAL: NCT01533025
Title: Single Bundle Anterior Cruciate Ligament Reconstruction in Active Young Men: Free Tendon Achilles Allograft vs. Bone-tendon Achilles Allograft
Brief Title: Single Bundle Anterior Cruciate Ligament Reconstruction in Active Young Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Police Hospital (Other Government)
Responsible Party: Principal Investigator, Jung Ho Noh, Principal Investigator, National Police Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NPH2008-007
Record Dates: First submitted 2012-02-10; First posted 2012-02-15 (Estimated); Last update posted 2012-02-15 (Estimated); Status verified 2012-02

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: anterior cruciate ligament; Achilles; free tendon; bone-tendon; free tendon Achilles allograft; Achilles allograft with calcaneal bone block on its end
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Anterior Cruciate Ligament Reconstruction

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bone-tendon Achilles allograft group (Active Comparator): the group which underwent anterior cruciate ligament reconstruction using bone-tendon Achilles allograft
  Interventions: Procedure: anterior cruciate ligament reconstruction
- free tendon Achilles allogarft group (Active Comparator): the group which underwent anterior cruciate ligament reconstruction using free tendon Achilles allograft
  Interventions: Procedure: anterior cruciate ligament reconstruction

INTERVENTIONS:
Procedure: anterior cruciate ligament reconstruction — single bundle anterior cruciate ligament reconstruction with Achilles allograft

SUMMARY:
The clinical outcomes of anterior cruciate ligament reconstruction using free tendon Achilles allograft are comparable to those using Achilles allograft with bone block on its end.

ELIGIBILITY:
Inclusion Criteria:

* male subjects
* subjects who had concomitant medial collateral ligament injury which was managed conservatively
* subjects who had meniscus tear which was managed by partial meniscectomy

Exclusion Criteria:

* subjects who underwent a subtotal or total meniscectomy, meniscal repair, or meniscal transplantation due to meniscus injury
* subjects who underwent an operation due to any concomitant ipsilateral ligament injuries
* subjects who underwent microfracture or cartilage transplantation due to full thickness cartilage injury
* female
* subjects who were older than 45
* subjects who had histories of injuries on either knee

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2008-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Lysholm score | 2 years

SECONDARY OUTCOMES:
side-to-side differences | 2 years
  the differences of anterior displacement of tibia under loading between normal knee and reconstructed knee

CONTACTS AND LOCATIONS:
Overall Officials: Jung Ho Noh, M.D., Ph.D., Principal Investigator — National Police Hospital
Locations (1):
- National Police Hospital, Seoul, South Korea